CLINICAL TRIAL: NCT00328666
Title: Cardiovascular Effects of Iyengar Yoga vs. Enhanced Usual Care in Patients With High-normal to Stage I Hypertension
Brief Title: The Penn Lifestyle Modification and Blood Pressure Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 802058 LIMBS; NIH grant number AT002353-02; NCT00271895 (obsolete NCT alias)
Record Dates: First submitted 2006-05-18; First posted 2006-05-22 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Behavioral: Iyengar yoga
Behavioral: Enhanced nutritional care classes

SUMMARY:
The purpose of this study is to compare the effects of 12 weeks of structured classes of either iyengar yoga (IY) or an enhanced usual care intervention on blood pressure, heart rate variability, quality of life measures, lipid measures, and safety in patients with high-normal to stage I hypertension.

DETAILED DESCRIPTION:
This is a single site, parallel, non-blinded, randomized controlled trial to assess the safety and efficacy of 12 weeks of structured IY vs. enhanced usual care in adults with high-normal to stage I HTN. All potential subjects will be screened first by telephone and then by an outpatient visit at the General Clinical Research Center (GCRC) at either the hospital of the University of Pennsylvania (HUP) or the Presbyterian Medical Center (PMC). Eligible subjects will then make 4 visits to the GCRC where, during 3 visits, they will be admitted overnight to have non-invasive 24 hour recordings of blood pressure and heart rate variability as well as periodic blood and urine collections. In order to assess durability of biologic effects once the formal intervention is stopped, we added a 4 week follow up visit. The entire study duration is 18 weeks (16 weeks post-randomization) and includes a total of 5 visits. Subjects will be randomized to either the IYP or Blood Pressure Education Program (BPEP) which will be incorporated into off-site, small group classes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing to, and have the capacity for, giving written informed consent.
* Between the ages of 18 and 70
* Blood pressure (BP) criteria: systolic blood pressure (SBP) of > 130 but < 160 mm Hg and diastolic blood pressure (DBP) < 100 mmHg
* All subjects must be willing to comply with all study-related procedures.

Exclusion Criteria:

* Female subjects who are pregnant or post partum < 3 months
* Subjects currently taking blood pressure lowering medications or dietary supplements (magnesium, potassium, calcium > 1200 mg/day, fish oils > 2000 mg/day, ephedra, hawthorn, forskolin)
* Non-dominant arm circumference > 50 cm
* Subjects with body mass index (BMI) >= 40.0 or < 18.5 kg/m2
* Subjects who have practiced IY in the last 12 months or those who have practiced any form of yoga > 2 times (2x)/month in the previous 6 months.
* Subjects who have received an experimental drug, used an experimental medical device within 30 days prior to screening, or who gave a blood donation of greater than or equal to one pint within 8 weeks prior to screening.
* Subjects with diabetes mellitus
* Subjects with established cardiovascular disease
* Subjects with known arrhythmias such as atrial flutter or fibrillation or those with cardiac pacemakers
* Current users (within the previous 30 days) of any tobacco products
* History of renal insufficiency based on estimated glomerular filtration rate < 60 ml/min
* Women who consume > 10 alcoholic drinks per week and men who consume > 15 drinks per week.
* Subjects with known autonomic neuropathy (e.g: Shy-Drager, orthostatic hypotension)
* Subjects with known secondary causes of hypertension (renal artery stenosis, pheochromocytoma, coarctation of aorta, hyperaldosteronemia)
* Regular use of benzodiazepines, anti-psychotic drugs or corticosteroids (> 1x per month). Stable doses (3 months) of antidepressants (selective serotonin reuptake inhibitors [SSRIs] or tricyclic antidepressants [TCAs]) will be allowed.
* Known severe musculoskeletal problems such as spinal stenosis that may limit participation in yoga
* Subjects who actively practice (> 2x/month) other mind-body therapy (MBT) such as Qigong, Tai Chi, or meditation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure

SECONDARY OUTCOMES:
heart rate variability
lipids
safety markers
quality of life measures
physiologic markers of stress
insulin resistance
pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Townsend, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States